CLINICAL TRIAL: NCT02270359
Title: Research on Infarction With Open Arteries Using OCT and CMR (RIO)
Brief Title: Research on Infarction With Open Arteries Using OCT and CMR
Acronym: RIO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1R01HL124204-01
Record Dates: First submitted 2014-10-01; First posted 2014-10-21 (Estimated); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; CAD
MeSH Terms: conditions — Myocardial Infarction | interventions — Contrast Media; Gadolinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MI without obstructive CAD (Other): MI without obstructive CAD, with OCT and CMR imaging
  Interventions: Device: OCT; Procedure: CMR; Drug: contrast agent, Gadolinium

INTERVENTIONS:
Device: OCT — Optical coherence tomography (OCT): Intracoronary imaging for amount and type of plaque as well as plaque rupture, ulceration, dissection and/or thrombosis.
Procedure: CMR — Cardiac magnetic resonance imaging (CMR): MRI of the heart to identify areas of infarction (damage) and/or edema (smelling)
Drug: contrast agent, Gadolinium — Gadolinium contrast will be administered during CMR

SUMMARY:
The purpose of this study is to determine the prevalence of plaque disruption and to assess the composition of disrupted plaques in patients with myocardial infarction (MI) and non-obstructive coronary artery disease (CAD) using optical coherence tomography (OCT). Additionally, cardiac magnetic resonance imaging (CMR) will be used to detect myocardial abnormalities, which will be correlated to OCT findings to gain insight into the mechanisms of MI in patients with non-obstructive coronary artery disease (i.e. "open arteries").

DETAILED DESCRIPTION:
In this single center, observational study, patients of both sexes with MI who are referred for cath will be enrolled. Those who have no obstructive CAD on clinically indicated coronary angiography, defined as no stenosis of >50% in any major epicardial vessel, will undergo coronary OCT just after the clinically indicated diagnostic angiogram, and CMR within 1 week, typically within 72-96 hours. Participants will be followed for clinical events for at least 1 year. 20 fully eligble participants will be recruited at NYU Langone Medical Center and Bellevue Hospital Center among a projected 200 enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic symptoms compatible with diagnosis of acute coronary syndrome (ACS) (chest pain or anginal equivalent symptoms at rest or new onset exertional anginal equivalent symptoms)
* Objective evidence of myocardial infarction (either or both of the following): Elevation of troponin to above the laboratory upper limit of normal (ULN) or ST segment elevation of ≥1mm on 2 contiguous ECG leads
* Willing to provide informed consent and comply with all aspects of the protocol
* Age ≥ 21 years

Exclusion Criteria:

* Stenosis ≥50% of any major epicardial vessel on invasive angiography, as determined by the angiographer at the time of clinically ordered cardiac cath.
* History of known obstructive CAD at angiography, including history of percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG)
* Recent use of vasospastic agents, such as cocaine, triptans, ergot alkaloids (≤1 month)
* Alternate explanation for troponin elevation, such as hypertensive urgency, acute exacerbation of heart failure, chronic elevation due to kidney disease, pulmonary embolism, cardiac trauma
* Coronary dissection apparent on angiography
* Excessive coronary tortuosity which, in the opinion of the angiographer, increases the risks of OCT
* eGFR<30 or contraindication to additional contrast needed for OCT in the opinion of the angiographer or treating physician
* Contraindication to MRI (including but not limited to MRI-incompatible metal implants or foreign bodies)
* Pregnancy
* Thrombolytic therapy for STEMI (qualifying event)

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
The prevalence of plaque disruption | 1 Week

SECONDARY OUTCOMES:
Prevalence and pattern of LGE and myocardial edema Prevalence of different plaque types according to OCT Proportion of patients with identifiable MI etiology based on study testing | 1 week

OTHER OUTCOMES:
Event rate in follow-up: death, MI, heart failure, stroke | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Harmony Reynolds, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States